CLINICAL TRIAL: NCT05906394
Title: A Pre-market, Open-label, Single-arm Study to Evaluate b.Bone for Posterolateral Fusion Treatment of Degenerative Thoracolumbar, Lumbar or Lumbosacral Spinal Disease.
Brief Title: A Pre-market Study to Evaluate b.Bone for Posterolateral Fusion (b.Spine Clinical Trial).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GreenBone Ortho S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-P010-0122; CIV-23-03-042713 (Other: EUDAMED Number)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Spinal Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posterolateral Fusion (Experimental): Patients recruited for clinical investigation will undergo up to a three-level posterolateral fusion (PLF) procedure with b.Bone granules.
  Interventions: Procedure: Posterolateral Fusion

INTERVENTIONS:
Procedure: Posterolateral Fusion — Posterolateral spinal fusion is a neurosurgical or orthopaedic surgical technique that joins two or more vertebrae. This procedure can be performed at any level in the spine (cervical, thoracic, lumbar, or sacral) and prevents any movement between the fused vertebrae.

SUMMARY:
Prospective, open-label, single-arm clinical investigation. The purpose of this clinical investigation is to evaluate the bone substitute b.Bone in posterolateral fusion treatment of degenerative thoracolumbar, lumbar or lumbosacral spinal conditions, in terms of performance and safety.

Subjects who meet the study selection will undergo up to a three-level posterolateral fusion using b.Bone in combination with autologous bone in a 1:1 ratio. Subjects will be followed up at discharge, week 6, Month 3, Month 6, and Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years old.
2. Patients requiring posterolateral fusion treatment for degenerative thoracolumbar, lumbar, or lumbosacral spinal conditions up to 8 levels.
3. Patients willing and able to attend the follow-up visits and procedures foreseen by the study protocol.
4. Patients who have provided written informed consent to participate in the study and the processing of personal data before any study procedure is performed.

Exclusion Criteria:

1. Any previous surgical attempt(s) for spinal fusion (revision surgery) of the intended segment(s).
2. Patients who have been treated with chemotherapy or radiotherapy within 12 months before the enrolment.
3. Indication for spinal fusion because of an acute traumatic reason, like a spinal fracture.
4. Bone infection.
5. Bone malignant tumor(s).
6. Concomitant infectious systemic diseases,
7. Inflammatory systemic diseases,
8. Concomitant myeloproliferative disorders,
9. Active autoimmune disease,
10. Known or suspected allergy or hypersensitivity to the b.Bone device components,
11. Calcium metabolism disorder (i.e. hypercalcemia),
12. Known hyperthyroidism or autonomous thyroid adenoma.
13. Patients currently treated with systemic immunosuppressive agents.
14. Patients who are currently enrolled in another clinical study that would directly interfere with the current study, except when the patient is participating in a purely observational registry with no associated treatments.
15. Body mass index (BMI) larger than 36 (morbidly obese).
16. Known severe osteoporosis.
17. Patients requiring instrumented fusion in the cervical spine.
18. Woman who is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Successful fusion rate by CT scan assessments after surgery. | 12 months

SECONDARY OUTCOMES:
Successful fusion rate by CT scan assessments after surgery. | 6 months
Back and Leg pain assessed by Visual Analog Scale. | Baseline, 6 weeks, 3, 6, and 12 months post-treatment.
Functional activity assessed by Oswestry Disability Index. | Baseline, 6 weeks, 3, 6, and 12 months post-treatment.
Quality of life assessed by Health Questionnaire | Baseline, 6 weeks, 3, 6, and 12 months post-treatment.
Neurological function | Baseline, 3, 6, and 12 months post-treatment.
  Maintenance/improvement of neurological function postoperatively versus baseline.
Rate of Adverse Events through the clinical trial period. | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbanti Bròdano, Dr, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli, Bologna - Italy
Locations (2):
- Klinikum Magdeburg, Magdeburg, Germany
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No